CLINICAL TRIAL: NCT06210997
Title: Factors Determining Time Allocation of a Multiple-Choice Question Examination: The Students' Perspective
Brief Title: Factors Determining Time Allocation of a MCQ Examination
Status: Completed | Type: Observational
Sponsor: Suranaree University of Technology (Other)
Responsible Party: Principal Investigator, CHATCHAI, Associate Professor Dr. Chatchai Kreepala, M.D., Suranaree University of Technology
Other Study IDs: EC-64-102
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Factors Determining Time Allocation of a Multiple-Choice Question Examination
Keywords: MCQ; medical assessment; medical education; testing time estimation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Questionaires — The questionnaire was done online by the participants from second to fifth-year medical students.

SUMMARY:
The MCQ is one of the objective assessment methods. It is proper to evaluate the cognitive domain of learners with high objectivity. However, there are no definite criteria for determining the appropriate exam time. The ability to comprehend the meaning of a text, when reading, cannot be directly applied to reading for decision-making or answering questions.

DETAILED DESCRIPTION:
The study was conducted at the Institute of Medicine, Suranaree University of Technology in Thailand. The research participants were second to fifth-year medical students who had taken MCQ tests during their preclinical and clinical years between the academic years 2021-2022. All examinations in this study were computer-based, closed book, single best answer MCQs written in English. The participants were Thai, non-native English speakers A questionnaire was chosen as the data collection method due to the ease of administering it to new fourth-year medical students with minimal disruption to their learning activities. Convenience sampling was used to randomly select second to fifth-year medical students as the students would not be identifiable. An online survey or questionnaire-based study was used to collect information from participants in this study. If the data was unsaturated, triangulation data from a group of interviews would consist of students from different rotations to receive as much information on students' perspectives as possible

ELIGIBILITY:
Inclusion Criteria:

* Medical students (2nd- 5th years) at Institute of Medicine, Suranaree University of Technology

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The research participants were both preclinical and clinical years of medical students between the academic years 2021-2022. In the preclinical years, the study included three organ systems (hematology, urinary, and gastrointestinal system). Meanwhile, six clinical learning subjects from two major departments, which were Medicine and Surgery, were included. The medical students from another academic year who were re-sitting for the examination in 2021-2022 were included.
Sampling Method: Non-Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Factors Determining Time Allocation of a Multiple-Choice Question Examination: The Students' Perspective | June 2021-SEP 2022
  The authors were interested in exploring the aspects of the medical students' perspective about the factors affecting their discission on MCQs answering

SECONDARY OUTCOMES:
Equation for Medical Multiple-Choice Question Testing Time Estimation | June 2021-SEP 2022
  The authors generated a specific computer program that integrated with the operating system of the examination. Technical specific features included the ability to calculate the speed of students taking MCQ exams with images or videos in the questions or options.

CONTACTS AND LOCATIONS:
Overall Officials: Chatchai Kreepala, M.D., Principal Investigator — Institute of Medicine, Suranaree University of Technology
Locations (1):
- Institute of Medicine, Suranaree University of Technology, Nakhon Ratchasima, Thailand

IPD SHARING:
Plan to Share IPD: No
the students' IDs were blind from origianal data